CLINICAL TRIAL: NCT06472856
Title: Vasomotor Symptom Alleviation Through Acupuncture in Patients With Prostate Cancer
Acronym: VASA Pro
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Bon Secours Hospital, Cork (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24017
Record Dates: First submitted 2024-06-12; First posted 2024-06-25 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acupuncture (Experimental)
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture will be given using single use sterile stainless steel 34 gauge (Japanese size: 0.20 X 30 mm) filoform needles. Skin will be swabbed with an alcohol prep pad before acupuncture is administered. Needles will be inserted 0.5 to 1.0 centimetres deep into the skin and gently manipulated to create the deqi sensation. No electrical stimulation will be used.

SUMMARY:
A pilot study to assess the acceptability and efficacy of acupuncture in alleviating vasomotor symptoms (hot flushes and night sweats) in Irish patients with prostate cancer receiving androgen deprivation therapy.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a histologically confirmed diagnosis of prostate cancer and currently be treated with androgen deprivation therapy with or without additional prostate cancer therapies.
* Patients under the care of a Medical Oncologist in either Bons Secours Hospital or Cork University Hospital
* All participants must be experiencing moderate to severe vasomotor symptoms as defined by a score of 4 or more on the Hot Flash Index.

Exclusion Criteria:

* Patients under 18.
* Patients with HFI scores below 4.
* Patients not currently being treated with androgen deprivation therapy.
* Patients with contraindications to acupuncture.
* Patients already receiving acupuncture for vasomotor symptoms.
* Patients unwilling to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention | Completed after 6 weeks of acupuncture sessions and repeated 3 months after acupuncture has finished
  Specially designed questionnaire

SECONDARY OUTCOMES:
Changes in symptom interference scores | Completed after 6 weeks of acupuncture sessions and repeated 3 months after acupuncture has finished
  Changes in the Hot Flash Related Daily Interference Scale (HFRDIS). The scale is measured from 0-10, with lower scores indicating a better outcomes
Changes in sleep quality | Completed after 6 weeks of acupuncture sessions and repeated 3 months after acupuncture has finished
  Changes in Pittsburgh Sleep Quality Index (PSQI). Each answer is rated between 0-3, and a higher global score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Bons Secours Hospital, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No